CLINICAL TRIAL: NCT02628106
Title: Lipo-prostaglandin E1 Improves Renal Hypoxia Evaluated by BOLD-MRI in Patients
Brief Title: Lipo-prostaglandin E1 Improves Renal Hypoxia Evaluated by BOLD-MRI in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhicheng Li, A graduate student, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOLD-1981
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Results first posted 2016-05-24 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Alprostadil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lipo-prostaglandin E1 (Experimental): all patients received 10 ug lipo-PGE1 intravenously once daily for consecutive 14 days.
  Interventions: Drug: Lipo-PGE1

INTERVENTIONS:
Drug: Lipo-PGE1 — all patients received 10 ug lipo-PGE1 intravenously once daily for consecutive 14 days
  Other Names: alprostadil

SUMMARY:
The purpose of this study is to evaluate the effect of lipo-prostaglandin E1 （lipo-PGE1) on renal oxygenation in patients with diabetic nephropathy by blood oxygenation level dependent magnetic resonance imaging (BOLD-MRI).patients with stable chronic kidney disease (CKD) were included. All patients were divided into two groups: diabetic nephropathy（DN) and CKD without diabetes. In addition to the conventional treatments, all patients received 10 ug lipo-PGE1 intravenously once daily for consecutive 14 days. Kidney BOLD-MRI were performed before and after lipo-PGE1 administration to acquire bilateral renal cortical R2*(CR2*) and medullary R2* (MR2*) values. Meanwhile, the clinical indexes at baseline and under lipo-PGE1 including 24 hours urinary protein and serum creatinine were collected. the investigators want to prove Lipo-PGE1 can improve kidney medullary oxygenation in patients with DN.

DETAILED DESCRIPTION:
R2* maps were calculated using the in-house software in Matlab (version 7.0, The MathWorks, Inc., Cambridge, MA, USA) on a pixel-by-pixel basis by fitting㏑(signal intensity) versus echo time. The R2* map was windowed from 0 to 60 s-1.

Regions of interest (ROIs) with unfixed size (7 to 53 pixels) were defined at the upper, middle and lower poles of both kidneys in the medulla and cortex in the renal hilum plane based on the anatomical images. Three ROIs were placed in the medulla and cortex, respectively, carefully avoiding vessels, renal sinus and susceptibility artifacts, yielding a total of 6 ROIs in both kidneys. The values in each ROI were averaged for the bilateral cortex and medulla. To prevent significant bias from measurement variability, each sample was measured independently by three professional radiologists with more than 5 years of experience who were blinded to the clinical results. Thereafter, assuming the tests were coincident, the results were the averaged.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic kidney disease

Exclusion Criteria:

* Intolerance to lipo-PGE1, contraindication for MRI, concurrent urinary tract infection, acute kidney injury, acute cardiovascular and cerebrovascular complications and diabetic emergencies, with the use of corticosteroid and diureses.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: fang liu, doctor, Study Chair — Department of Nephrology, West China Hospital of Sichuan University
Locations (1):
- Zhichengli, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our overall recruiting cycle for 40 days, mainly for patients with chronic kidney disease patients, which is divided into diabetic nephropathy and non-diabetic patients
Pre-assignment Details: Chronic kidney disease patients were divided into diabetic nephropathy and non-diabetic group, ordinary chronic kidney disease patients with diabetes mellitus were excluded
Groups:
- Diabetic Nephropathy,Chronic Kidney Disease: all patients receivedlipo-prostaglandin E1,10ug per day, iv for 14 consecutive days.renal hypoxia in patients with diabetic nephropathy was improves evaluate via blood oxygenation level dependent magnetic resonance imaging
Period: Overall Study
Arm/Group | Diabetic Nephropathy,Chronic Kidney Disease
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: age > 18 years
Arm/Group | Lipo-prostaglandin E1
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — All applicable patients with CKD were eligible for this study. Other inclusion criteria were as follows: an age > 18 years and a diagnosis of type 2 diabetes based on the definition of the World Health Organization
  years | 59 (13)
Gender [Count of Participants; unit: Participants] — men and women randomly, but try to match proportion
  Participants
    Female | 12
    Male | 9
Region of Enrollment [Number; unit: participants] — A random sample, west China hospital, in accord with a standard 21 people
  participants
    China | 21
R2* values [Mean (Standard Deviation); unit: 1/ms] — Deoxyhemoglobin, as an endogenous contrast agent, is paramagnetic; the change in deoxyhemoglobin level can cause inhomogeneity in the magnetic field in the local tissue. R2* is a measure of the tissue content of deoxyhemoglobin, which is inversely proportional to the oxygen content in tissue. Thus, a decrease in R2* implies decreased deoxyhemoglobin concentrations and increased oxygen content in tissue.
  1/ms | 23.32 (6.48)

OUTCOME MEASURES:

1. Primary Outcome: the Change of Tissue Content of Deoxyhemoglobin Assessed by BOLD-MRI
Description: the R2* value at the time after 14days of lipo-PGE1 intravenously minus the value at the baseline，R2* is a measure of the tissue content of deoxyhemoglobin. Which is inversely proportional to oxygen content in tissue
Time Frame: baseline and after 14days of lipo-PGE1 intravenously
Population: A random sample, west China hospital, in accord with a standard 21 people,age > 18 years
Measure: Mean (Standard Deviation); unit: 1/ms
Groups:
- Diabetic Nephropathy,Chronic Kidney Disease: all patients received lipo-prostaglandin E1,10ug per day, iv for 14 consecutive days.renal hypoxia in patients with diabetic nephropathy was improves evaluate via blood oxygenation level dependent magnetic resonance imaging
Arm/Group | Diabetic Nephropathy,Chronic Kidney Disease
Number analyzed (Participants) | 21
1/ms | 22.04 (6.15)

ADVERSE EVENTS:
Time Frame: 1 year
Description: We assessed the 21 participants, but none of the participants had serious Adverse Event
Arm/Group | Diabetic Nephropathy,Chronic Kidney Disease
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
the small study population and absence of a placebo group and healthy volunteers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No